CLINICAL TRIAL: NCT06351709
Title: Acute Effects of Heat, Cold and Stretching on Knee Proprioception and Vertical Jump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Umut Paksoy, lecturer, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A47
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: proprioception; vertical jump; heat; streching; cold pack

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hot Pack Group (Experimental): Hot pack application was applied to the participants in the hot group to warm the extremities locally after the pre-tests were completed. For the application of hotpack, which is a superficial and moist temperature agent, a Chattanooga ® brand hotpack pad (DJO Global, Chattanooga; CA, USA) with 10 slices and a size of 28 cm x 39 cm was used. The hotpack pad was taken with the help of tongs from the Chattanooga ® brand hot pack boiler (DJO Global, Chattanooga; CA, USA) at 80° temperature and wrapped in a total of 5 layers with the help of 2 towels. A hotpackpad was placed on each knee of the participant. Hotpack pads were applied for 15 minutes in total.
  Interventions: Other: Hot pack application
- Cold Pack Group (Experimental): For participants in the cold group, MSD ® brand cold pack gel (MVS Inmotion, MSD cold pack; Weftdijk 1502830, Belgium), 15 cm x 25 cm in size, was used to cool the extremities locally. The cold pack gel, kept in the freezer, was wrapped in a paper towel and placed on the knee area. Cold pack was applied to both knees for a total of 15 minutes.
  Interventions: Other: Cold pack application
- Stretching Group (Experimental): Static stretching technique was applied to the quadriceps and hamstring muscle groups in both the dominant and non-dominant extremities of the participants in the stretching group. All stretches were performed twice for 20 seconds with a 3-second rest.
  Interventions: Other: Stretching
- Control Group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Other: Stretching — Static stretching technique was applied to the quadriceps and hamstring muscle groups in both the dominant and non-dominant extremities of the participants in the stretching group. All stretches were performed twice for 20 seconds with a 3-second rest.
  Arms: Stretching Group
Other: Hot pack application — Hot pack application was applied to the participants in the hot group to warm the extremities locally after the pre-tests were completed. For the application of hotpack, which is a superficial and moist temperature agent, a Chattanooga ® brand hotpack pad (DJO Global, Chattanooga; CA, USA) with 10 slices and a size of 28 cm x 39 cm was used. The hotpack pad was taken with the help of tongs from the Chattanooga ® brand hot pack boiler (DJO Global, Chattanooga; CA, USA) at 80° temperature and wrapped in a total of 5 layers with the help of 2 towels. A hotpackpad was placed on each knee of the participant. Hotpack pads were applied for 15 minutes in total.
  Arms: Hot Pack Group
Other: Cold pack application — For participants in the cold group, MSD ® brand cold pack gel (MVS Inmotion, MSD cold pack; Weftdijk 1502830, Belgium), 15 cm x 25 cm in size, was used to cool the extremities locally. The cold pack gel, kept in the freezer, was wrapped in a paper towel and placed on the knee area. Cold pack was applied to both knees for a total of 15 minutes.
  Arms: Cold Pack Group

SUMMARY:
The aim of our study is to investigate the effects of heat, cold and stretching on knee proprioception and vertical jump. 60 healthy individuals were randomized into hot, cold, stretching and control groups of 15 each. Pre-test and post-test measurements were made immediately after the application. Knee proprioception was measured with a digital goniometer using the EPD (joint position sense) test. Vertical jump heights were measured with contact mat by countermovement (CMJ) and squat splash (SQS) tests.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* Agreeing to participate in the study and being informed Approving the Volunteer Consent Form

Exclusion Criteria:

* Having a history of surgery in the knee area
* Movement in lower extremity joints that may affect measurements have limitations.
* Having vision, hearing and balance impairment.
* May cause peripheral neuropathy and deep sensory loss, or loss of proprioception may be caused by other mechanisms having diseases.
* Have a neurological or systemic disease that affects balance and coordination have.
* Describing very severe pain in any part of the lower extremity.
* Being pregnant.
* Having cognitive dysfunction, lack of cooperation
* Having any disease that may cause inability to dry

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Distance Measurement | Before and immediately after application
  Two types of vertical jump distances, squat jump and countermovement jump, were evaluated using a Fusion Sport ® brand jump meter (Fusion Sport, SmartJump; Colorado, USA) with a sensitivity of 1 nanometer, which is one thousandth of an antimeter. Both tests were repeated a total of 3 times and the best results were recorded.
Joint Position Sense Measurement | Before and immediately after application
  For the active joint position sense test, which measures the individual's ability to find the taught target angle, a BASELINE ® brand digital goniometer (BASELINE ® Evaluation Instruments, Digital Absolute + Axis goniometer; NY, USA) with a sensitivity of 0.1° was used.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipan Tıp Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No